CLINICAL TRIAL: NCT06971055
Title: Evaluation of Antimicrobial Efficacy of Moringa Oleifera Leaf Extract Versus Sodium Hypochlorite as Root Canal Irrigants in Pulpectomy of Nonvital Primary Molars: A Randomized Clinical Trial
Brief Title: Moringa Oleifera vs Sodium Hypochlorite for Root Canal Irrigation in Nonvital Primary Molars
Acronym: MORvNAOCL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alawi Taha A Alaidarous, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Moringa vs Sodium Hypochlorite
Record Dates: First submitted 2025-05-02; First posted 2025-05-14 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Dental Caries; Pulp Necrosis; Primary Tooth Pulpectomy; Pediatric Dentistry; Endodontic Infection
Keywords: Moringa oleifera; Sodium hypochlorite; Root canal irrigants; Pulpectomy; Primary molars; Enterococcus faecalis; Antimicrobial efficacy; Pediatric endodontics; Coagulase-Negative Staphylococci
MeSH Terms: conditions — Dental Caries; Dental Pulp Necrosis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Hypochlorite Group (Experimental): Participants in this group will receive root canal irrigation using sodium hypochlorite during pulpectomy of nonvital primary molars. A 3 mL solution will be used per canal following standard clinical procedures.
  Interventions: Drug: Sodium hypochlorite
- Moringa oleifera Leaf Extract Group (Experimental): extract of Moringa oleifera leaves prepared as a solution, used as a natural antimicrobial root canal irrigant.
  Interventions: Biological: Moringa Oleifera Leaf Extract

INTERVENTIONS:
Drug: Sodium hypochlorite — sodium hypochlorite solution will be used as a root canal irrigant during pulpectomy in primary molars. A volume of 3 mL will be delivered into each canal using a syringe with a side-vented needle. Irrigation will be followed by microbial sampling for blood agar
  Arms: Sodium Hypochlorite Group
Biological: Moringa Oleifera Leaf Extract — extract of Moringa oleifera leaves will be used as an intracanal irrigant during pulpectomy. A volume of 3 mL will be used per canal, and post-irrigation microbial samples will be analyzed using the same methods as the control group.
  Arms: Moringa oleifera Leaf Extract Group

SUMMARY:
This randomized clinical trial aims to evaluate and compare the antimicrobial efficacy of Moringa Oleifera leaf extract versus sodium hypochlorite as root canal irrigants in pulpectomy of nonvital primary molars in pediatric patients. The study will assess bacterial reduction using blood agar

DETAILED DESCRIPTION:
This randomized clinical trial is designed to compare the antimicrobial efficacy of Moringa Oleifera leaf extract and sodium hypochlorite when used as root canal irrigants in the pulpectomy of nonvital primary molars in children aged 4 to 7 years. Root canal disinfection in pediatric endodontics is essential due to the complex anatomy of primary teeth and the potential systemic implications of untreated infections.

Sodium hypochlorite (NaOCl) is widely used due to its strong antimicrobial and tissue-dissolving properties but is associated with cytotoxic effects and safety concerns in children. Moringa Oleifera, a plant rich in bioactive compounds such as flavonoids and isothiocyanates, has demonstrated antimicrobial, anti-inflammatory, and antioxidant properties, offering a potentially safer and natural alternative.

A total of 38 participants will be randomly assigned to two equal groups. Group 1 will receive root canal irrigation with 2.5% NaOCl, while Group 2 will be irrigated using an ethanol extract of Moringa Oleifera leaves. The primary outcome will be the diameter of the inhibition zone against Coagulase-Negative Staphylococci measured using a blood agar. The secondary outcome will be the diameter of the inhibition zone against Enterococcus Faecalis measured using a blood agar

The study will be conducted at the outpatient clinics of the Pediatric Dentistry and Dental Public Health Department at the Faculty of Dentistry, Cairo University. All procedures will be performed by a single operator (the principal investigator) using a standardized protocol. Data collection will be blinded at the laboratory and statistical analysis levels to minimize bias.

The results of this study aim to determine whether Moringa Oleifera extract can be a safe, effective, and biocompatible alternative to sodium hypochlorite in pediatric root canal irrigation, ultimately enhancing clinical outcomes and patient experience

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 7 years
* Clinically and radiographically diagnosed with nonvital primary molars requiring pulpectomy
* Cooperative children who can undergo dental treatment
* Healthy-appearing children with no systemic, physical, or mental disorders

Exclusion Criteria:

* Medically compromised or uncooperative children
* Primary molars indicated for extraction due to:
* Advanced root resorption (more than two-thirds)
* Teeth near exfoliation
* Deep subgingival caries preventing proper restoration
* Excessive mobility (Miller's Grade 2 or higher)

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Zone of inhibition against Coagulase-Negative Staphylococci | "Day 1 (Pre- and post-irrigation samples collected during the same visit)"
  "Primary Outcome: The antimicrobial efficacy of both types of irrigants... based on the diameter of the zone of inhibition

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No